CLINICAL TRIAL: NCT01898728
Title: Comparison of the Effectiveness of Povidone-iodine in Reducing Conjunctival Bacterial Load Prior to Cataract Surgery in Patients Treated With a Lidocaine Gel Dilating Formulation Versus Eye Drops: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lidocaine gel vs drops
Record Dates: First submitted 2013-07-07; First posted 2013-07-12 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2013-07

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — Gels

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liquid preoperative medications (Active Comparator): Liquid preoperative medications
  Interventions: Drug: topical povidone-iodine after premedication with topical liquid eye drops
- Gel preoperative medications (Active Comparator): Gel preoperative medications
  Interventions: Drug: topical povidone-iodine after premedication with topical gel

INTERVENTIONS:
Drug: topical povidone-iodine after premedication with topical liquid eye drops
  Arms: Liquid preoperative medications
Drug: topical povidone-iodine after premedication with topical gel
  Arms: Gel preoperative medications

SUMMARY:
The eye contains a lens that focuses light. A clouding of the lens is known as a cataract. Cataracts decrease vision. The treatment for cataracts is cataract surgery. Cataract surgery is one of the most commonly performed surgical procedures. Although rare, complications of cataract surgery are significant given the number of people who have surgery each year and more serious complications may have a significant impact on the vision and quality of patients. Endophthalmitis is an infection in the eye and it is one of the worst complications of cataract surgery. Most of these infections are caused by bacteria from the patient's skin and conjunctiva, which makes cleaning the skin and eye before surgery very important. Before cataract surgery, patients receive an umber of eye drops; many surgical centers have a combination of medications in a thick gel, so that the medications remain in the eye for a long period of time, which may improve their effect. Laboratory studies suggest that the antibacterial effect of cleaning solutions may be inhibited by gels but this has not been proven, and many believe it to be untrue. This study is to compare the amount of bacteria on the eye prior to surgery in patients receiving a gel formulation of the medications before surgery as compared to those receiving the same medication in eye drop (liquid) form.

DETAILED DESCRIPTION:
The human eye contains a crystalline lens that focuses light onto the retina. A clouding of the lens is known as a cataract. Cataracts progressively decrease visual acuity and contrast sensitivity. Cataracts are the leading cause of blindness worldwide. The current standard of practice for treating cataracts is cataract extraction using phacoemulsification, an ultrasound technology to liquefy and aspirate the lens material, and the implantation of an intraocular lens (IOL) to clearly refocus light onto the retina. Cataract surgery is one of the most commonly performed surgical procedures. Although rare, complications of cataract surgery are significant given the number of people who have surgery each year and more serious complications may have a significant impact on the vision and quality of life of patients.

Endophthalmitis is an intraocular inflammation involving both the anterior and posterior segments of the eye attributable to bacterial or fungal pathogens. Postoperative endophthalmitis is one of the most devastating complications of cataract surgery and despite aggressive treatment, only approximately half of patients achieve better than 20/40 vision and many patients remain no light perception (NLP). The majority of causative organisms are from the patient's skin and conjunctival flora, making preoperative reduction in conjunctival flora a key component of endophthalmitis prophylaxis. The Endophthalmitis Vitrectomy Study (EVS) revealed that 70% of infections are due to coagulase-negative Staphylococcus, 9.9% due to Staphylococcus aureus, 2.2% from Enterococcus, and 5.9% from Gram-negative bacteria. A recent systematic review evidenced a postoperative endophthalmitis rate of 0.265% from 2000 to 2003, compared with 0.087% in the previous decade. There are numerous theories to the increase in incidence, including a move to topical anaesthesia and change in wound construction techniques. It is difficult for prospective studies to be detect differences in the rate of endophthalmitis as the incidence is low. Currently, only topical povidone-iodine and intracameral antibiotics (cefuroxime, vancomycin, and moxifloxacin) have been shown to decrease the rate of endophthalmitis.

Prior to cataract surgery while in the preoperative area, patients receive a number of eye drops, frequently including antibiotics, corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), anaesthetics and mydriatics/cycloplegics. Many surgical centres, including the Regional Eye Institute at the St. Joseph's Centre for Ambulatory Care have a pharmacy-prepared combination of the above medications in a viscous gel, such that the medications remain on the ocular surface for a prolonged period of time thus enhancing efficacy.

Topical lidocaine gel is an anaesthetic that is used prior to cataract surgery in many institutions.Studies demonstrating that the antiseptic effect of topical povidone-iodine may be inhibited by topical lidocaine gel have been published. Boden et al. performed a basic science study inoculating culture media with bacteria and then exposing them to topical lidocaine gel, topical povidone-iodine or topical povidone-iodine after lidocaine gel. Their results revealed that the antiseptic effect of povidone-iodine was inhibited by previous treatment with lidocaine gel. Moreover, a retrospective observational case series found that 2 of 7 cases of postoperative endophthalmitis occurred after topical lidocaine gel use. Most recently, Doshi et al. in the laboratory setting confirmed the inhibitory effect of lidocaine gel prior to povidone-iodine and also revealed that if povidone-iodine was applied prior to lidocaine gel, the iodine was able to act as an antiseptic as usual.

The previous studies reveal that there may be an inhibition of the antiseptic effect of povidone-iodine when topical lidocaine gel is applied first in the laboratory setting. This has not been shown clinically.

ELIGIBILITY:
Inclusion Criteria

* Aged greater than 18 years
* Able to give informed consent
* Undergoing uncomplicated cataract surgery

Exclusion Criteria

* Hypersensitivity to any of the components of the premedication
* Hypersensitivity to povidone-iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The number of Colony Forming Units (CFUs) | Period before surgery

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton King Campus, Hamilton, Ontario, Canada